CLINICAL TRIAL: NCT04346186
Title: COVID-19: Investigation of Transmission and Immunisation Among Hospital Staff
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Nordsjaellands Hospital (Other); Hvidovre University Hospital (Other); Rigshospitalet, Denmark (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Kasper Iversen, Professor, Herlev Hospital
Other Study IDs: RegHCOVIDScreening
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital Staff in the Capital Region of Denmark
  Interventions: Diagnostic Test: IgM and IgG diagnostic kits to SARS-CoV-2; Diagnostic Test: Elisa-test for IgM and IgG to SARS-CoV-2
- Healthy volunteer blood donors
  Interventions: Diagnostic Test: IgM and IgG diagnostic kits to SARS-CoV-2; Diagnostic Test: Elisa-test for IgM and IgG to SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: IgM and IgG diagnostic kits to SARS-CoV-2 — Diagnostic kits for IgM/IgG antibodies to SARS-CoV-2
Diagnostic Test: Elisa-test for IgM and IgG to SARS-CoV-2 — Elisa-test for IgM and IgG to SARS-CoV-2

SUMMARY:
During the COVID-19 pandemic several countries have seen a high risk of transmission for health care personnel, with some countries having as many 20-25% of nurses and doctors either infected or showing symptoms of COVID-19.

In this prospective cohort study, we will systematically screen all hospital staff in the Capital Region of Denmark for IgM and IgG antibodies against SARS-CoV-2 using a point of care tests and an Elisa kit.

Testing will be offered 3 times: In April 2020, Maj 2020 and September 2020. All participants will submit a questionnaire regarding exposures, risk factors and symptoms of COVID-19 in relation to each testing. Follow-up will be through electronic patient records and national registries.

We will compare the group of health care personnel with data from a control group of healthy volunteer blood donors from the Danish Blood Donor Study.

The aim of the study is to investigate the proportion of hospital staff with SARS-CoV-2 antibodies during the study period compared to a control group representing the Danish population. We will compare the test characteristics of the two methods of testing, a point of care test and Elisa.

Further, we will investigate the extent to which prior immunization or infection is protective for future infection with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Consent to participation
* Employed at a Hospital in the Capitial Region of Denmark

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All staff with any form of contact with patients, employed at any hospital in the Capital Region of Denmark will be offered to participate at their place of employment.
Sampling Method: Non-Probability Sample
Enrollment: 44698 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Positive IgM/IgG tests | At inclusion
  Proportion of hospital staff who have a positive IgM/IgG tests for antibodies to SARS-CoV-2 on point of care test and/or Elisa compared to the background population
Positive IgM/IgG tests | 1 month
  Proportion of hospital staff who have a positive IgM/IgG tests for antibodies to SARS-CoV-2 on point of care test and/or Elisa compared to the background population
Positive IgM/IgG tests | 5 month
  Proportion of hospital staff who have a positive IgM/IgG tests for antibodies to SARS-CoV-2 on point of care test and/or Elisa compared to the background population
Comparison of the point of care test and Elisa | At inclusion
  Comparison of the resultat from the point of care test and with results from Elisa
Comparison of the point of care test and Elisa | 1 months
  Comparison of the resultat from the point of care test and with results from Elisa
Comparison of the point of care test and Elisa | 5 months
  Comparison of the resultat from the point of care test and with results from Elisa
Re-infection rate | 180 days
  Number of patients, who were tested positive for antibodies on an earlier test and later are infected with COVID-19
Re-infection rate | 360 days
  Number of patients, who were tested positive for antibodies on an earlier test and later are infected with COVID-19
IgM/IgG positive participants on follow-up test | 1 month
  Proportion of IgM/IgG positive participants with a lasting immune response. This will be the participants who are still positive on follow-up
IgM/IgG positive participants on follow-up test | 5 months
  Proportion of IgM/IgG positive participants with a lasting immune response. This will be the participants who are still positive on follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Iversen, Prof., Principal Investigator — Herlev-Gentofte Hospital; Henning Bundgaard, Prof., Principal Investigator — Rigshospitalet, Denmark; Henrik Ullum, Prof., Principal Investigator — Rigshospitalet, Denmark; Thomas Benfield, Prof., Principal Investigator — Hvidovre University Hospital; Susanne Dam Poulsen, Prof., Principal Investigator — Rigshospitalet, Denmark; Jørgen Rungby, Prof., Principal Investigator — Bispebjerg Hospital; Fredrik Folke, Associate prof., Principal Investigator — Akutberedskabet; Thea Kølsen Fischer, Principal Investigator — Nordsjaellands Hospital; Ove Andersen, Prof., Principal Investigator — Hvidovre University Hospital; Ida Hageman, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (14):
- Denmark (14):
  - Herlev Hospital, Herlev, Capital Region
  - Bispebjerg Hospital, København NV, Capital Region
  - Psykiatrisk Center Ballerup, Ballerup Municipality
  - Psykiatrisk Center København, Copenhagen
  - Rigshospitalet, Copenhagen
  - Psykiatrisk Center Amager, Copenhagen
  - Psykiatrisk Center Stolpegaard, Gentofte Municipality
  - Børne- og Ungdomspsykiatrisk Center, Glostrup Municipality
  - Psykiatrisk Center Glostrup, Glostrup Municipality
  - Nordsjaellands Hospital, Hillerød
  - Psykiatrisk Center Nordsjælland, Hillerød
  - Psykiatrisk Center Sankt Hans, Roskilde
  - Bornholms Hospital, Rønne
  - Psykiatrisk Center Bornholm, Rønne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iversen K, Kristensen JH, Hasselbalch RB, Pries-Heje M, Nielsen PB, Knudsen AD, Fogh K, Norsk JB, Andersen O, Fischer TK, Juul Jensen CA, Torp-Pedersen C, Rungby J, Ditlev SB, Hageman I, Mogelvang R, Gybel-Brask M, Dessau RB, Sorensen E, Harritshoj L, Folke F, Sten C, Engel Moller ME, Benfield T, Ullum H, Jorgensen CS, Erikstrup C, Ostrowski SR, Nielsen SD, Bundgaard H. Seroprevalence of SARS-CoV-2 antibodies and reduced risk of reinfection through 6 months: a Danish observational cohort study of 44 000 healthcare workers. Clin Microbiol Infect. 2022 May;28(5):710-717. doi: 10.1016/j.cmi.2021.09.005. Epub 2021 Sep 17. PMID 34543759
- [Derived] Iversen K, Bundgaard H, Hasselbalch RB, Kristensen JH, Nielsen PB, Pries-Heje M, Knudsen AD, Christensen CE, Fogh K, Norsk JB, Andersen O, Fischer TK, Jensen CAJ, Larsen M, Torp-Pedersen C, Rungby J, Ditlev SB, Hageman I, Mogelvang R, Hother CE, Gybel-Brask M, Sorensen E, Harritshoj L, Folke F, Sten C, Benfield T, Nielsen SD, Ullum H. Risk of COVID-19 in health-care workers in Denmark: an observational cohort study. Lancet Infect Dis. 2020 Dec;20(12):1401-1408. doi: 10.1016/S1473-3099(20)30589-2. Epub 2020 Aug 3. PMID 32758438